CLINICAL TRIAL: NCT06740448
Title: Investigating the Effects of Green Tea on Whole Blood Viscosity
Brief Title: Investigating the Effects of Green Tea on Blood Viscosity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other); Royal Berkshire NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: UREC 24/22
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Disease
Keywords: Flavanol; Green Tea; Blood Viscosity; Older Adults
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Tea

STUDY DESIGN:
Intervention Model Description: A randomised, single blind, crossover design with a 3 week washout period between conditions investigating the acute effects (over 2 and 8 hours) of green tea on blood viscosity
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Green Tea (Experimental): 200 mL green tea on first visit
  Interventions: Dietary Supplement: Green Tea; Dietary Supplement: Control (Hot Water)
- Hot Water (Placebo Comparator): 200 mL hot water on first visit
  Interventions: Dietary Supplement: Green Tea; Dietary Supplement: Control (Hot Water)

INTERVENTIONS:
Dietary Supplement: Green Tea — 200 mL Green Tea
Dietary Supplement: Control (Hot Water) — 200 mL hot water

SUMMARY:
A diet high in flavonoids is becoming more established as beneficial to human health. Recent data suggest that the regular consumption of flavanols can reduce the numbers of deaths by cardiovascular disease at a population level. The mechanisms for these reductions in deaths by cardiovascular disease are still debated and little is known about their impacts on factors affecting blood viscosity. The metabolism of flavanols is complex, with different metabolites being predominant in the blood at different time points. Therefore, in this study, we will investigate the effects of green tea, a well-known source of flavanols, on blood viscosity at different time points. This will be assessed in healthy individuals with no history of cardiovascular disease aged 65+ years old. Blood viscosity will be measured before, and 2hours and 8hours after the consumption of green tea.

DETAILED DESCRIPTION:
Participants will first be screened via a questionnaire on RedCap. This will include a list of exclusion and inclusion criteria. Examples of what will be included are: must be a non-smoker, no history of CVD or CVD in immediate family, no history of metabolic diseases, no food allergies, or intolerances and not be on any medication for cardiovascular purposes (e.g. aspirin or blood pressure medication).

Before confirmation, a screening visit will be undertaken where checks for regular haematocrit, blood pressure, plasma triglycerides, blood glucose and inflammatory markers and BMI will be taken. This will involve a 4.5 ml blood sample. Additionally, the research nurse will assess the potential participant's veins, and participants who do not have 2 'good' veins for giving blood will be excluded from the trial.

Following recruitment, participants will be asked to follow a set of criteria for the 24 hours prior to participating in the study. This will include, following a low polyphenol diet and not consuming any over the counter medication, caffeine or alcohol for 24 hours prior to participating. Participants will also be asked to attend fasted for 12 hours. Participants will also be asked to not take part in any vigorous/aerobic exercise in the 24 hours leading up to the study.

Following recruitment, and on arrival, participants will be asked to confirm they have followed the requirements for the previous 24 hours and full informed consent will be obtained from the participant. Participants will complete a spot urine test to measure osmolality as a measure of hydration. Participants will be asked to sit in a rested position for 15 min prior to each blood sample. Blood pressure will then be measured followed by a blood sample (17.5ml). The blood sample will be passed through the viscometer to assess whole blood and plasma viscosity and part of the blood sample will be used to measure haematocrit, inflammatory markers and blood lipids. The participant will then be given 200 mL green tea. They will be asked to consume this within 15 minutes. The intervention will be provided in an opaque cup with a lid on and the participant will be asked not to remove the lid so that the contents is not revealed to them. This will be followed by a low flavonoid breakfast. The same blood sample and urine test will then be taken at 2 hours and 8 hours after the start of consuming the drink, and these will be processed in the same way. A low flavonoid meal will also be provided between the 2- and 8-hour blood sample. A second visit will involve the exact same protocol; however, the participants will be given hot water as a control condition.

On the first of two visits, the participant will be asked to fill out a food frequency questionnaire. The order of green tea/control visits will be randomised and counterbalanced. In the 12-hours leading up to the visit, participants will be asked to consume 500 mL of water (a bottle will be provided). Throughout the visit, participants will be provided with unlimited water to drink and the total volume that has been consumed between each blood sample throughout the study will be recorded. On the second visit, the participant will be asked to replicate this amount.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 65 years and older
* Non-smoker Participants with at least 2 'good' veins for giving blood

Exclusion Criteria:

* Participants under (BMI <18.5 kg/m2) or extremely over-nourished (BMI >30 kg/m2)
* Participants on prescription medication for CVD or regularly taking blood thinning drugs such as aspirin.
* Participants with a history of CVD or CVD in immediate family/ high resting blood pressure
* Participants with any food allergies/intolerances
* Participants with a history of metabolic diseases/ high resting blood glucose
* Participants with high resting levels of inflammatory markers (CRP)
* Participants on hormone replacement therapy
* Participants with abnormal red blood cell count or low haemoglobin stores

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Whole Blood Viscosity | Baseline to 2 hours and 8 hours

SECONDARY OUTCOMES:
Plasma Viscosity | Baseline to 2 hours and 8 hours
Blood Triglycerides | Baseline to 2 hours and 8 hours
C-reactive protein | Baseline to 2 hours and 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hugh Sinclaire Unit of Human Nutrition, Departmeant of Food and Nutrition, University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes